CLINICAL TRIAL: NCT05735990
Title: Retrospective Clinical Investigation of the Safety and Performance of 640PM Trifocal IOL Implantation in Patients With Cataract and/or Ametropia (Hyperopia, Myopia) and/or Presbyopia
Status: Completed | Type: Observational
Sponsor: Medicontur Medical Engineering Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: M_640PM_ES_2202
Record Dates: First submitted 2022-10-28; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cataract; Presbyopia; Hyperopia; Myopia; Pseudophakia
MeSH Terms: conditions — Cataract; Presbyopia; Hyperopia; Myopia; Pseudophakia | interventions — Lenses, Intraocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 640PM implanted: Patients implanted binocularly with Medicontur's intraocular lens model 640PM.
  Interventions: Device: Intraocular lens

INTERVENTIONS:
Device: Intraocular lens — Aspheric hydrophilic acrylic IOL for implantation into the capsular bag

SUMMARY:
The clinical investigation objective is to evaluate safety and performance outcomes of trifocal IOL implantation to improve vision in patients with cataract and/or ametropia (hyperopia, myopia) and/or presbyopia.

Retrospective data from preoperative status up to 12 month postoperative status will be collected from patients that were implanted with Medicontur's 640PM intraocular lens:

* Preoperative status: Preoperative Screening and Baseline
* Surgery: IOL implantation
* M1: 1 month +/- 2 weeks postoperative follow-up
* M3: 3 months +/- 1 month postoperative follow-up
* M12: 12 months +/- 3 months postoperative follow-up

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females above 18 years of age;
* Pseudophakic patients implanted with 640PM IOLs (Medicontur Medical Engineering Ltd. Inc., Zsámbék, Hungary);
* Diagnosis of cataract and/or ametropia and/or presbyopia;
* Subject who provided express consent authorizing the use of medical record data for biomedical research purposes. Patients who have participated in at least two follow up visits in the 12 months following IOL implantation
* Patients for which the retrospective data for the primary endpoint is available and at least half of all the secondary endpoints measured in the time ranges specified in the protocol.

Exclusion Criteria:

* Patients with any eye condition that could affect vision (corneal ectasia, retinal diseases, glaucoma, uveitis, dry eye or amblyopia, etc.);
* regular anterior corneal astigmatism ≥ 1.20 D or irregular astigmatism ≥ 0.5 μm measured with Pentacam at 4 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 years old and older) with cataract and/or ametropia (hyperopia, myopia) and/or presbyopia, who has binocular 640PM IOL implantation.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Corrected distance visual acuity (CDVA); | 12 months after IOL implantation

SECONDARY OUTCOMES:
visual acuity at all intended distances (UDVA; CDVA, UIVA, DCIVA, UNVA, DCNVA) | 1 and 12 months after IOL implantation;
Manifest spherical equivalent refraction (SEQ) | 3 and 12 months after IOL implantation
VADC (monocular with best distance correction) under photopic conditions | 3 months after IOL implantation
CSDC (monocular with best distance correction): To evaluate CSDC under photopic conditions | 3 months after IOL implantation;
CSDC (binocular without best distance correction) under photopic and mesopic conditions | 12 months after IOL implantation;
Visual Function by VF-14 | 12 months after IOL implantation;
Patient satisfaction self-reported by the participant | 12 months after IOL implantation
Visual disturbances (photic phenomena, dysphotopsia) self-reported by the participant | 12 months after IOL implantation
spectacle independence self-reported by the participant | 12 months after IOL implantation

OTHER OUTCOMES:
Secondary surgical intervention rate | 12 months after IOL implantation;
Collect and evaluate ocurrence of adverse events detected | from surgery to 12 months after IOL implantation
PCO rate | 12 months after IOL implantation
Nd-YAG capsulotomy rate | 12 months after IOL implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vithas Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez J, Srinivasan S, Burguera N, Martinez J, Rodriguez-Vallejo M. One-year follow-up of a multifocal intraocular lens with optimized elevated phase shift. J Cataract Refract Surg. 2023 Oct 1;49(10):1018-1024. doi: 10.1097/j.jcrs.0000000000001266. PMID 37464551